CLINICAL TRIAL: NCT03236441
Title: Biochemical and Reno-protective Effects of Remote Ischemic Pre-conditioning on Contrast-induced Acute Kidney Injury
Brief Title: Biochemical Effects of Remote Ischemic Pre-Conditioning on Contrast-induced Acute Kidney Injury
Acronym: BRICK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oladipupo Olafiranye, MD, MS (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Oladipupo Olafiranye, MD, MS, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19090247; 1R21DK113486-01A1 (NIH)
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Contrast-induced Acute Kidney Injury
Keywords: remote ischemic conditioning; contrast-induced nephropathy; cardiac catheterization; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RIPC Group (Active Comparator): 3 cycles of blood pressure cuff inflations to occlusive pressure of 200 mmHg for 5 minutes and deflation for 5 minutes
  Interventions: Device: RIPC
- Sham-RIPC Group (Sham Comparator): 3 cycles of blood pressure cuff inflations to non-occlusive pressure of 10 mmHg for 5 minutes and deflation for 5 minutes (Control)
  Interventions: Device: Sham-RIPC

INTERVENTIONS:
Device: RIPC — Remote ischemic preconditioning
  Arms: RIPC Group
Device: Sham-RIPC — Control
  Arms: Sham-RIPC Group

SUMMARY:
This a prospective, double-blind, sham-controlled, randomized clinical trial to study the effects of remote ischemic preconditioning on acute kidney injury, vascular and renal biomarkers in patients with non-ST elevation myocardial infarction and unstable angina undergoing coronary angiography and/or percutaneous coronary intervention.

DETAILED DESCRIPTION:
The BRICK study is a prospective, double-blind, sham-controlled, randomized clinical trial in patients with non-ST elevation myocardial infarction and unstable angina undergoing coronary angiography and/or percutaneous coronary intervention who are at high risk for acute kidney injury. The study will investigate the effects of remote ischemic preconditioning before cardiac catheterization on rate of acute kidney injury and novel biomarkers of renal injury/protection within 48hrs of coronary angiography and/or percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-ST elevation myocardial infarction or unstable angina
* Referral for cardiac catheterization and percutaneous coronary intervention
* Contrast-induced acute kidney injury risk score of ≥11

Exclusion Criteria:

* Inability to give informed consent
* unstable blood pressure (systolic blood pressure > 200 or <90 mmHg)
* History of allergy to contrast media
* Peripheral vascular disease of upper limb
* Renal disease requiring dialysis
* Placement of arteriovenous fistula and arteriovenous graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oladipupo Olafiranye, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olafiranye O, Straub AC, Zhang Y, Chaudhary R, Miller MP, Trivedi K, Hoang L, Khalifa O, Ladejobi A, Thoma FW, Feng N, Rahman A, Kellum JA; BRICK Trial Investigators. Remote Ischemic Preconditioning Prevents Acute Kidney Injury Following Coronary Angiography: The BRICK Randomized Clinical Trial. JACC Adv. 2025 Sep;4(9):102092. doi: 10.1016/j.jacadv.2025.102092. Epub 2025 Aug 23. PMID 40850057

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 110 patients enrolled in this study, 1 patient withdrew after signing informed consent and prior to randomization. As a result, a total of 109 patients were randomized or assigned to RIPC or Sham-RIPC groups.
Period: Overall Study
Arm/Group | RIPC Group | Sham-RIPC Group
Started | 54 | 55
Completed | 54 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Predominantly elderly patients with unstable angina and non-ST elevation myocardial infarction undergoing coronary angiography with high modified Mehran risk score for acute kidney injury were enrolled in this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | RIPC Group | Sham-RIPC Group | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76 [71 to 82] | 75 [71 to 80] | 75 [71 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 45 | 47 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 50 | 51 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Acute Kidney Injury
Description: acute kidney injury is defined as a relative increase in serum creatinine of ≥ 0.3mg/dl within 48 hours post catheterization compared with baseline creatinine before coronary angiography.
Time Frame: 24-48 hours post coronary angiography
Population: 54 patients in the RIPC group and 55 patients in the sham-RIPC group were included in the primary outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC Group | Sham-RIPC Group
Number analyzed (Participants) | 54 | 55
Participants | 8 | 16

2. Secondary Outcome: The Product of Urinary (Tissue Inhibitor of Metalloproteinases 2) X (Insulin-like Growth Factor-binding Protein 7)
Description: Novel renal biomarker. The product of urinary tissue inhibitor of metalloproteinases 2 and insulin-like growth factor-binding protein 7 is measured and reported as a single test in (ng/ml)2/1000 unit. Higher value in general indicates higher risk of acute kidney injury. The range is between 0.3 and 10.
Time Frame: 0-48hrs
Measure: Mean (Standard Deviation); unit: (ng/ml)2/1000
Arm/Group | RIPC Group | Sham-RIPC Group
Number analyzed (Participants) | 54 | 55
(ng/ml)2/1000
  Baseline | 0.39 (0.51) | 0.51 (0.51)
  Post RIPC/Sham-RIPC | 0.71 (1.58) | .49 (.56)
  24hrs post coronary angiography | 0.67 (0.66) | 0.67 (0.89)
  48hrs post coronary angiography | 0.68 (0.66) | 0.89 (0.84)

3. Secondary Outcome: Number of Patients With Major Adverse Cardiovascular and Cerebrovascular Event
Description: Composite outcome including rehospitalization for myocardial infarction, hospitalization for heart failure, repeat revascularization, stroke, and cardiac death.
Time Frame: 6 months post coronary angiography
Population: Patients with unstable angina and non-ST segment elevation myocardial infarction at high risk for acute kidney injury referred for coronary angiography and or percutaneous coronary angiography.
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC Group | Sham-RIPC Group
Number analyzed (Participants) | 54 | 55
Participants | 9 | 20

4. Secondary Outcome: Number of Patients With Major Adverse Kidney Event
Description: Composite outcome including persistent renal impairment, use of renal replacement therapy, and all-cause death.
Time Frame: 6 months post coronary angiography.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC Group | Sham-RIPC Group
Number analyzed (Participants) | 54 | 55
Participants | 4 | 6

5. Secondary Outcome: Cyclic Guanylate Monophosphate (cGMP) Level
Description: Higher level of cyclic guanylate monophosphate is associated with greater vessel dilatation and blood flow. Cyclic GMP was measured in nanomolar (nM).
Time Frame: 0-48 Hrs
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | RIPC Group | Sham-RIPC Group
Number analyzed (Participants) | 54 | 55
nM
  Baseline | 60.12 (84.71) | 55.19 (147.46)
  Post RIPC | 68.28 (112.56) | 59.66 (181.04)
  24 Hours post coronary angiogram | 62.91 (89.36) | 55.22 (116.02)
  48 Hours post coronary angiogram | 65.61 (96.01) | 45.04 (65.00)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | RIPC Group | Sham-RIPC Group
All-Cause Mortality (participants affected / at risk) | 4/54 | 4/55
Serious Adverse Events (participants affected / at risk) | 4/54 | 8/55
Other Adverse Events (participants affected / at risk) | 5/54 | 14/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIPC Group (N=54) | Sham-RIPC Group (N=55)
Repeat Coronary Revascularization (Cardiac disorders) | 4 | 6
Stroke (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RIPC Group (N=54) | Sham-RIPC Group (N=55)
Major adverse cardiovascular and cerebrovascular events (Cardiac disorders) | 5 | 14
Major Adverse Kidney Events (Renal and urinary disorders) | 4 | 6

LIMITATIONS AND CAVEATS:
The population studied was predominantly elderly male patients with non-ST elevation myocardial infarction or unstable angina.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03236441/Prot_SAP_001.pdf